CLINICAL TRIAL: NCT02172040
Title: A Prospective Randomized Placebo Controlled Study to Evaluate the Effect of Celecoxib on the Efficacy and Safety of Amlodipine in Subjects With Hypertension Requiring Antihypertensive Therapy
Brief Title: Study to Evaluate the Effect of Celecoxib on the Efficacy and Safety of Amlodipine in Subjects With Hypertension Requiring Antihypertensive Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kitov Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Organization: KitovPharma (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KIT-302-03-01; 2013-005381-19 (EudraCT Number)
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
Keywords: High blood pressure; Systolic blood pressure; Diastolic blood pressure; Antihypertensive
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Amlodipine+Celecoxib (Experimental): Over-encapsulated 10 mg amlodipine besylate tablet + over-encapsulated 200 mg celecoxib capsule once a day for two weeks
  Interventions: Drug: Over-encapsulated 10 mg amlodipine besylate tablet; Drug: Over-encapsulated 200 mg celecoxib capsule
- Amlodipine+Placebo (Active Comparator): Over-encapsulated 10 mg amlodipine besylate tablet + matched placebo capsule for over-encapsulated celecoxib capsule once a day for two weeks
  Interventions: Drug: Over-encapsulated 10 mg amlodipine besylate tablet; Drug: Matched placebo capsule for over-encapsulated celecoxib capsule
- Placebo+Celecoxib (Placebo Comparator): Matched placebo capsule for over-encapsulated amlodipine besylate tablet + over-encapsulated 200 mg celecoxib capsule once a day for two weeks
  Interventions: Drug: Over-encapsulated 200 mg celecoxib capsule; Drug: Matched placebo capsule for over-encapsulated amlodipine besylate tablet
- Placebo+Placebo (Sham Comparator): Matched placebo capsule for over-encapsulated amlodipine besylate tablet + matched placebo capsule for over-encapsulated celecoxib capsule once a day for two weeks
  Interventions: Drug: Matched placebo capsule for over-encapsulated celecoxib capsule; Drug: Matched placebo capsule for over-encapsulated amlodipine besylate tablet

INTERVENTIONS:
Drug: Over-encapsulated 10 mg amlodipine besylate tablet — Over-encapsulated 10 mg amlodipine besylate tablet once a day for two weeks
  Other Names: Norvasc
  Arms: Amlodipine+Celecoxib; Amlodipine+Placebo
Drug: Matched placebo capsule for over-encapsulated celecoxib capsule — Matched placebo capsule for over-encapsulated celecoxib capsule once a day for two weeks
  Other Names: Placebo
  Arms: Amlodipine+Placebo; Placebo+Placebo
Drug: Over-encapsulated 200 mg celecoxib capsule — Over-encapsulated 200 mg celecoxib capsule once a day for two weeks
  Other Names: Celebrex
  Arms: Amlodipine+Celecoxib; Placebo+Celecoxib
Drug: Matched placebo capsule for over-encapsulated amlodipine besylate tablet — Matched placebo capsule for over-encapsulated amlodipine besylate tablet once a day for two weeks
  Other Names: Placebo
  Arms: Placebo+Celecoxib; Placebo+Placebo

SUMMARY:
The purpose of this study was to evaluate the effect of celecoxib on the efficacy and safety of amlodipine besylate in subjects with newly diagnosed hypertension requiring antihypertensive therapy.

This study was conducted to support a future marketing application for KIT-302. Kitov Pharma Ltd. (Kitov) is developing KIT-302, an oral fixed combination drug product (FCDP) consisting of the calcium channel blocker amlodipine besylate and the nonsteroidal anti-inflammatory drug (NSAID) celecoxib, as a "convenience reformulation" FCDP to facilitate and improve patient compliance with the once a day (qd) administration of its individual components, amlodipine and celecoxib.

The formulation of KIT-302 consists of amlodipine besylate and celecoxib co-formulated in a single immediate release tablet. However, for this study, two separate capsules were utilized: one containing a commercial celecoxib capsule (Celebrex®) or matched placebo capsule and one containing a commercial amlodipine besylate tablet (Norvasc®) or matched placebo tablet.

The study hypothesis was that treatment with the amlodipine besylate containing capsule plus the celecoxib containing capsule would reduce blood pressure (BP) in subjects with hypertension with an efficacy that is not substantially inferior to the effect of amlodipine besylate alone (i.e., the amlodipine containing capsule plus the matched placebo for the celecoxib capsule).

The United States (US) Food and Drug Administration (FDA) recently approved KIT-302, under the brand name Consensi® (amlodipine and celecoxib) tablets [New Drug Application (NDA) 210045] for the following indication: "patients for whom treatment with amlodipine for hypertension and celecoxib for osteoarthritis are appropriate. Lowering blood pressure reduces the risk of fatal and nonfatal cardiovascular events, primarily strokes and myocardial infarctions."

ELIGIBILITY:
Inclusion Criteria:

1. Adult 40 to 75 years of age
2. Newly diagnosed hypertension that requires chronic pharmacological therapy. Specifically, the subject must meet both of the following criteria:

   1. Resting systolic BP ≥140 mmHg and ≤179 mmHg (where resting is defined as supine for at least 10 minutes with minimal interaction) at Initial Screening Visit
   2. SBPday >135 mmHg at Baseline Visit (Day 0)
3. Body Mass Index of 18.5 to 34.9 kg/m2
4. Healthy (other than hypertension) as determined by the Investigator based on medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests
5. A negative pregnancy test at Screening
6. Both males and women of child bearing potential agree to use adequate contraceptive methods while on study (from Screening through final study visit)
7. Able to comprehend and sign an informed consent form

Exclusion Criteria:

1. Resting systolic BP >179 mmHg or a resting diastolic BP >110 mmHg at Screening (where resting is defined as supine for at least 10 minutes with minimal interaction) or SBP24h >169 mmHg or DBP24h >110 mmHg at randomization
2. SBPday ≤135 mmHg at baseline (Day 0)
3. Weight <55 kg
4. Fragile health
5. Evidence of clinically significant findings on screening evaluations (clinical, laboratory, and ECG) which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of safety data
6. Current or recent history (within 4 weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection
7. Current clinically significant viral infection
8. History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin
9. Major surgery within 4 weeks prior to Screening
10. Presence of a malabsorption syndrome possibly affecting drug absorption (e.g., Crohn's disease or chronic pancreatitis)
11. Active peptic ulceration or history of gastrointestinal bleeding
12. History of myocardial infarction, congestive heart failure, or stroke
13. Any current cardiovascular disease
14. History of psychotic disorder
15. History of alcoholism or drug addiction or current alcohol or drug use that, in the opinion of the Investigator, will interfere with the subject's ability to comply with the dosing schedule and study evaluations
16. History of any illicit drug use within one year prior to Screening
17. Positive drug screen at Screening. A positive drug screen for opiates only (with all other drug tests negative) will not be a basis for exclusion if the subject took over-the-counter narcotics as indicated on the product label within 24 hours prior to the drug screen
18. Current treatment or treatment within 30 days prior to first dose of study drugs with another investigational drug or current enrollment in another clinical trial
19. Current treatment or treatment within 30 days prior to first dose of study drugs with an NSAID or systemic corticosteroid
20. Known history of human immunodeficiency virus, hepatitis B, or hepatitis C
21. Known hypersensitivity to amlodipine or celecoxib
22. Known hypersensitivity to the inactive ingredients in the over-encapsulated study drugs
23. Asthma, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria or other allergic type reactions after taking acetylsalicylic acid or NSAIDs including cyclooxygenase-2 inhibitors
24. Subjects who, in the opinion of the Investigator, are unable or unlikely to comply with the dosing schedule and study evaluations
25. Pregnant or lactating
26. Unable to correctly use ambulatory blood pressure monitor after instruction on its use
27. Subjects with Child-Pugh Class B or C cirrhosis;
28. Subjects currently taking a calcium channel blocker for any reason including angina. Subjects will not be withdrawn from these drugs to be enrolled in the trial
29. Creatinine clearance <50 ml/min as estimated by the Cockroft-Gault equation
30. Known cytochrome P450 2C9 poor metabolizer
31. Subjects with allergy or hypersensitivity to sulfonamides

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2015-11-19 (Actual); Study Completion 2015-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Paul Waymack, MD, ScD, Study Director — Kitov Pharma Ltd; Brendan Colgan, MD, Principal Investigator — Celerion; Claire Kightley, MB, Principal Investigator — Reading Clinical Research Aspect; David Collier, MBBS, PhD, BSc, Principal Investigator — Barts Health NHS Trust, William Harvey Heart Centre, Barts & The London, Queen Mary School of Medicine and Dentistry, Queen Mary, University of London; Paul Ivan, MBBS, Principal Investigator — Synexus Merseyside Clinical Research Centre; Veronika Horvathova, MD, Principal Investigator — Synexus Scotland Clinical Research Centre; Amit Mathew, MS, MBBS, Principal Investigator — Synexus Midlands Clinical Research Centre; Alexander Thompson, MB, BS, DRCOG, Principal Investigator — Reading Clinical Research Aspect; Mohamed Okily, MB, Principal Investigator — Synexus Manchester Clinical Research Centre; Richard Gaunt, MB, ChB, MRCGP, DRCOG, Principal Investigator — Rowden Surgery; Patrick Eavis, MBBS, DRCOG, DFFP, MRCGP, Principal Investigator — Oldfield Surgery; Arjun Ravi, MBBS, MRCP, Principal Investigator — The Medicines Evaluation Unit Ltd.
Locations (10):
- United Kingdom (10):
  - Celerion, Belfast, Antrim
  - The Medicines Evaluation Unit Ltd., Manchester, Greater Manchester
  - Reading Clinical Research Aspect, Ledbury, Herefordshire
  - Synexus Merseyside Clinical Research Centre, Liverpool, Merseyside
  - Oldfield Surgery, Bath, North East Somerset
  - Rowden Surgery, Chippenham, Wiltshire
  - Synexus Midlands Clinical Research Centre, Birmingham
  - Synexus Scotland Clinical Research Centre, Glasgow
  - Barts Health NHS Trust, William Harvey Heart Centre, Barts & The London, Queen Mary School of Medicine and Dentistry, Queen Mary, University of London, London
  - Reading Clinical Research Aspect, Reading

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent assessments to determine eligibility at the Initial Screening Visit (Day -7 to -2; 458 participants), Final Screening Visit (Day -1; 228 participants), and the morning prior to randomization (Study Day 0; 227 participants). A total of 306 participants were screen failures and the remaining 152 were randomized.
Groups:
- Placebo+Celecoxib: Matched placebo tablet for over-encapsulated amlodipine besylate tablet + over-encapsulated 200 mg celecoxib capsule once a day for two weeks
  Over-encapsulated 200 mg celecoxib capsule: Over-encapsulated 200 mg celecoxib capsule once a day for two weeks
  Matched placebo tablet for over-encapsulated amlodipine besylate tablet: Matched placebo tablet for over-encapsulated amlodipine besylate tablet once a day for two weeks
- Placebo+Placebo: Matched placebo tablet for over-encapsulated amlodipine besylate tablet + matched placebo capsule for over-encapsulated celecoxib capsule once a day for two weeks
  Matched placebo capsule for over-encapsulated celecoxib capsule: Matched placebo capsule for over-encapsulated celecoxib capsule once a day for two weeks
  Matched placebo tablet for over-encapsulated amlodipine besylate tablet: Matched placebo tablet for over-encapsulated amlodipine besylate tablet once a day for two weeks
Period: Overall Study
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Started | 49 | 45 | 31 | 27
Completed | 49 | 42 | 29 | 26
Not Completed | 0 | 3 | 2 | 1
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Not available for Day 13 & 14 visits | 0 | 0 | 1 | 0
Not completed — Family emergency abroad | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo | Total
Number analyzed (Participants) | 49 | 45 | 31 | 27 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.0) | 57.3 (9.4) | 54.9 (8.2) | 52.5 (9.1) | 56.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 10 | 10 | 56
  Male | 32 | 26 | 21 | 17 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 0 | 3
  White | 46 | 43 | 29 | 26 | 144
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 49 | 45 | 31 | 27 | 152
Average Daytime (9:00 to 21:00) Ambulatory Systolic Blood Pressure (SBPday) [Mean (Standard Deviation); unit: mmHg] | 148.7 (7.4) | 147.6 (8.7) | 150.8 (8.9) | 147.3 (8.6) | 148.5 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Average Daytime (9:00 to 21:00) Ambulatory Systolic Blood Pressure (SBPday) - Primary Endpoint
Time Frame: Baseline and 2 weeks
Population: Intent-to-treat (ITT): All randomized participants who received at least 1 dose of study drug and had at least a valid baseline ambulatory blood pressure monitor measurement (ABPM) and either: a) a valid Day 13-14 ABPM, where participant completed treatment or b) a valid Day 6-7 or Day 0-1 ABPM, where participant was withdrawn early.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 30 | 26
mmHg | -10.6 (9.2) | -8.83 (8.13) | -0.5 (8.8) | -2.11 (8.2)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; A serial gatekeeping strategy was used for the primary efficacy endpoint analysis. The primary comparison was a two-sample t-test to test the one-sided hypothesis that treatment with amlodipine + celecoxib was non-inferior to half of the effect achieved with amlodipine; Test type: Non-Inferiority — Non-inferiority margin definition: lower limit of the 95% confidence interval (CI) for amlodipine + celecoxib arm did not cross the 50% value for the amlodipine arm; p = 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Placebo+Celecoxib vs Placebo+Placebo; A serial gatekeeping strategy was used for the primary efficacy endpoint analysis. The secondary comparison was a two-sample t-test to test the one-sided hypothesis that treatment with placebo was superior to treatment with celecoxib. This was only to be performed if statistical significance was achieved for the primary comparison; Test type: Superiority; p = 0.491, t-test, 1 sided

2. Primary Outcome: Frequency of Adverse Events (Number of Participants Affected/Number of Participants at Risk)
Description: Including any untoward medical occurrence in a participant administered study drug, which do not necessarily have a causal relationship with the study drug [i.e., any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not related to the study drug].
Time Frame: 1 month
Population: Safety population: all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 31 | 27
Participants | 27 | 28 | 14 | 10
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo vs Placebo+Celecoxib vs Placebo+Placebo; Test type: Other; p = 0.166, Chi-squared

3. Secondary Outcome: Mean Change in Average 24-hour Ambulatory Systolic Blood Pressure (SBP24h)
Time Frame: Baseline and 2 weeks
Population: ITT population as described for primary outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 30 | 26
mmHg | -10.3 (8.9) | -8.02 (7.6) | -0.5 (7.8) | -1.19 (5.87)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Superiority; p = 0.177, t-test, 1 sided
Statistical Analysis 2: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Amlodipine+Celecoxib vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Amlodipine+Placebo vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 5: Comparison: Amlodipine+Placebo vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 6: Comparison: Placebo+Celecoxib vs Placebo+Placebo; Test type: Superiority; p = 0.719, t-test, 1 sided

4. Secondary Outcome: Mean Change in Average Night-time (01:00 to 06:00) Ambulatory Systolic Blood Pressure (SBPnight)
Time Frame: Baseline and 2 weeks
Population: ITT Population as described for primary outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 30 | 26
mmHg | -10.5 (10.6) | -6.35 (11.35) | -1.7 (12.3) | -1.42 (9.15)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Superiority; p = 0.069, t-test, 1 sided
Statistical Analysis 2: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Superiority; p = 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Amlodipine+Celecoxib vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Amlodipine+Placebo vs Placebo+Celecoxib; Test type: Superiority; p = 0.097, t-test, 1 sided
Statistical Analysis 5: Comparison: Amlodipine+Placebo vs Placebo+Placebo; Test type: Superiority; p = 0.064, t-test, 1 sided
Statistical Analysis 6: Comparison: Placebo+Celecoxib vs Placebo+Placebo; Test type: Superiority; p = 0.924, t-test, 1 sided

5. Secondary Outcome: Mean Change in Average 24-hour Ambulatory Diastolic Blood Pressure (DBP24h)
Time Frame: Baseline and 2 weeks
Population: ITT Population as described for primary outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 30 | 26
mmHg | -7.1 (5.6) | -4.8 (4.83) | -0.5 (4.6) | 0.22 (4.28)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Superiority; p = 0.038, t-test, 1 sided
Statistical Analysis 2: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Amlodipine+Celecoxib vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Amlodipine+Placebo vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 5: Comparison: Amlodipine+Placebo vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 6: Comparison: Placebo+Celecoxib vs Placebo+Placebo; Test type: Superiority; p = 0.562, t-test, 1 sided

6. Secondary Outcome: Mean Change in Average Daytime (9:00 to 21:00) Ambulatory Diastolic Blood Pressure (DBPday)
Time Frame: Baseline and 2 weeks
Population: ITT Population as described for primary outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 30 | 26
mmHg | -7.5 (6.4) | -5.53 (5.06) | -1.5 (5.6) | -0.32 (5.39)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Superiority; p = 0.104, t-test, 1 sided
Statistical Analysis 2: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Amlodipine+Celecoxib vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Amlodipine+Placebo vs Placebo+Celecoxib; Test type: Superiority; p = 0.002, t-test, 1 sided
Statistical Analysis 5: Comparison: Amlodipine+Placebo vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 6: Comparison: Placebo+Celecoxib vs Placebo+Placebo; Test type: Superiority; p = 0.419, t-test, 1 sided

7. Secondary Outcome: Mean Change in Average Night-time (01:00 to 06:00) Ambulatory Diastolic Blood Pressure (DBPnight)
Time Frame: Baseline and 2 weeks
Population: ITT Population as defined for primary outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 30 | 26
mmHg | -7.0 (8.6) | -3.23 (7.79) | 0.3 (7.1) | 0.01 (6.23)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Superiority; p = 0.028, t-test, 1 sided
Statistical Analysis 2: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Amlodipine+Celecoxib vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Amlodipine+Placebo vs Placebo+Celecoxib; Test type: Superiority; p = 0.051, t-test, 1 sided
Statistical Analysis 5: Comparison: Amlodipine+Placebo vs Placebo+Placebo; Test type: Superiority; p = 0.074, t-test, 1 sided
Statistical Analysis 6: Comparison: Placebo+Celecoxib vs Placebo+Placebo; Test type: Superiority; p = 0.878, t-test, 1 sided

8. Secondary Outcome: Mean Non-transformed Amlodipine Plasma Concentration
Time Frame: 24 hours post-dose on Day 14
Population: Pharmacokinetic (PK) population: subset of overall trial population, consisting of participants at Investigational sites capable of obtaining PK blood samples in a protected light environment. No amlodipine PK statistical analyses were performed for the PK participants in the placebo+celecoxib and placebo+placebo arms.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 24 | 20
pg/mL | 15,800.83 (4,161.929) | 23,453 (5,746.337)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Other; p < 0.001, t-test, 1 sided

9. Secondary Outcome: Mean Non-transformed Celecoxib Plasma Concentration
Time Frame: 24 hours post-dose on Day 14
Population: PK population: subset of overall trial population, consisting of participants at Investigational sites capable of obtaining PK blood samples in a protected light environment. No celecoxib PK statistical analyses were performed for the PK participants in the amlodipine+placebo and placebo+placebo arms.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amlodipine+Celecoxib | Placebo+Celecoxib
Number analyzed (Participants) | 24 | 15
ng/mL | 139.708 (86.504) | 138.667 (118.811)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Other; p = 0.977, t-test, 1 sided

10. Secondary Outcome: Mean Log-transformed Amlodipine Plasma Concentration
Time Frame: 24 hours post-dose on Day 14
Population: PK population: subset of overall trial population, consisting of participants at Investigational sites capable of obtaining PK blood samples in a protected light environment. No amlodipine PK statistical analyses were performed for the PK participants in the placebo+celecoxib and placebo+placebo arms.
Measure: Mean (Standard Deviation); unit: log(pg/mL)
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo
Number analyzed (Participants) | 24 | 20
log(pg/mL) | 9.634 (0.268) | 10.025 (0.310)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Amlodipine+Placebo; Test type: Other; p < 0.001, t-test, 1 sided

11. Secondary Outcome: Mean Log-transformed Celecoxib Plasma Concentration
Time Frame: 24 hours post-dose on Day 14
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: log(ng/mL)
Arm/Group | Amlodipine+Celecoxib | Placebo+Celecoxib
Number analyzed (Participants) | 24 | 15
log(ng/mL) | 4.785 (0.564) | 4.636 (0.781)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Other; p = 0.527, t-test, 1 sided

12. Secondary Outcome: Mean Change in Average Daytime (9:00 to 21:00) Ambulatory Systolic Blood Pressure (SBPday) - Secondary Endpoint
Time Frame: Baseline and 2 weeks
Population: ITT Population as described for primary outcome
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
Number analyzed (Participants) | 49 | 45 | 30 | 26
mmHg | -10.6 (9.2) | -8.83 (8.13) | -0.5 (8.8) | -2.11 (8.2)
Statistical Analysis 1: Comparison: Amlodipine+Celecoxib vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Amlodipine+Celecoxib vs Placebo+Placebo; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Amlodipine+Placebo vs Placebo+Celecoxib; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Amlodipine+Placebo vs Placebo+Placebo; Test type: Superiority; p = 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Amlodipine+Celecoxib | Amlodipine+Placebo | Placebo+Celecoxib | Placebo+Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/45 | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/45 | 0/31 | 0/27
Other Adverse Events (participants affected / at risk) | 17/49 | 17/45 | 5/31 | 6/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine+Celecoxib (N=49) | Amlodipine+Placebo (N=45) | Placebo+Celecoxib (N=31) | Placebo+Placebo (N=27)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 7 (8) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 6 (10) | 2 (3) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days